CLINICAL TRIAL: NCT04289194
Title: Phase 1/2 Clinical Study to Assess the Feasibility, Safety, Tolerability and Preliminary Efficacy of the Administration of HCR040, Allogeneic Adipose-derived Adult Mesenchymal Stem Cells, in Acute Respiratory Distress Syndrome
Brief Title: Clinical Study to Assess the Safety and Preliminary Efficacy of HCR040 in Acute Respiratory Distress Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Histocell, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALICELL-CT-01; 2019-002688-89 (EudraCT Number)
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2022-02

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; mesenchymal stem cells; anti-inflammation; allogenic; ARDS; acute lung injury; cell therapy
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — Clinical Trials, Phase I as Topic; Heart Rate; Clinical Trials, Phase II as Topic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HCR040 (Phase 1) (Experimental): Participants with moderate to severe acute respiratory distress syndrome (6 patients)
  Interventions: Drug: HCR040 (Phase 1)
- Control group (Phase 2) (Placebo Comparator): Participants with moderate to severe acute respiratory distress syndrome (10 patients)
  Interventions: Drug: Placebo (Phase 2)
- HCR040 (Phase 2) (Experimental): Participants with moderate to severe acute respiratory distress syndrome (10 patients)
  Interventions: Drug: HCR040 (Phase 2)

INTERVENTIONS:
Drug: HCR040 (Phase 1) — (Phase 1) Intravenous administration. Open label dose escalation, 3 patients in cohort 1 (1 million cells/kg) and 3 patients in cohort 2 (2 million cells/kg)
  Other Names: Allogeneic adipose-derived adult mesenchymal stem cells expanded and pulsed with H2O2
  Arms: HCR040 (Phase 1)
Drug: Placebo (Phase 2) — (Phase 2) Intravenous administration of vehicle solution
  Other Names: Saline solution
  Arms: Control group (Phase 2)
Drug: HCR040 (Phase 2) — (Phase 2) Intravenous administration of the maximum tolerated dose (1 million cells/kg or 2 million cells/kg)
  Other Names: Allogeneic adipose-derived adult mesenchymal stem cells expanded and pulsed with H2O2
  Arms: HCR040 (Phase 2)

SUMMARY:
The main objective of the study is to assess the feasibility, safety, and tolerability of the administration of HCR040, a drug whose active substance is HC016, allogeneic adipose-derived adult mesenchymal stem cells expanded and pulsed with H2O2, in patients with acute respiratory distress syndrome.

DETAILED DESCRIPTION:
HCR040 is an investigational medicinal product whose active substance is HC016, allogeneic adipose-derived adult mesenchymal stem cells expanded and pulsed with H2O2.

The main purpose of this study is to evaluate the safety and tolerability of a single administration of HCR040 using: a) two sequential escalating doses administered 96 hours post-injury to participants with moderate to severe acute respiratory distress syndrome (ARDS); and b) the determined maximum tolerated dose administered 96 hours post-injury to participants with moderate to severe ARDS. The study also includes initial exploration of efficacy.

Treatment is administered by intravenous injection.

The study has been divided into two phases:

Phase 1 (open label): 6 participants with moderate to severe ARDS will be included in 2 sequential cohorts.

Phase 2 (randomized, controlled, double-blind): 20 participants with moderate to severe ARDS will be randomly divided into two groups (control and treated).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years
* Patients with criteria of moderate to severe ARDS according to the Berlin Conference.
* Berlin criteria of moderate to severe ARDS given simultaneously during the 24 hours prior to entry into the study
* Patients with invasive mechanical ventilation in controlled mode (VC, PC or VCRP) adjusted to Vt≤8 mL/kg, Ppl <30 cmH2O and minimum PEEP of 8 cmH2O

Exclusion Criteria:

* Participation in a previous clinical study within 28 days prior to the ARDS situation
* Administration of a previous cell therapy product in the 5 years prior to this ARDS clinical situation
* Inability to obtain Informed Consent
* Hemodynamic instability that contraindicates the intravenous cellular administration, within the defined time frame for inclusion in the study
* Alveolar hemorrhage or hemoptysis
* LTSV situation (Limitation of life support treatments)
* Major trauma in the previous 5 days
* Neoplastic processes at any time
* EPOC or severe home asthma or any other type of chronic respiratory disease requiring respiratory oxygen
* Known Child-Pugh liver disease score > B9
* Pregnant women or women of childbearing age who are not using an adequate method of contraception, or who, if they are using it, are not willing to continue using it for the duration of the trial. If the patient is menopausal or sterile, it must be documented in the medical record
* Women who are breastfeeding if unwillingly to stop at the time of recruitment
* Pulmonary transplant
* Known grade III or IV pulmonary hypertension
* States of hypercoagulability
* History of DVP or PE in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
Number of adverse events as a measure of safety and tolerability of a single dose of HCR040 when administered by intravenous injection | One year

SECONDARY OUTCOMES:
Average stay in the Intensive Care Unit (ICU) 28 days after the administration of HCR040 | Day 28
Sequential Organ Failure Assessment (SOFA) index at 3, 7, 14, 21, and 28 days after the administration of HCR040 | Day 28
  SOFA index from 0 to 4 where lower scores represent improvement
Mechanical ventilation-free days 28 days after the administration of HCR040 | Day 28
Percent mortality 28 days after the administration of HCR040 | Day 28
Daily pulmonary mechanics values (Ppl, DP, CRS) | One year
Determination of lung damage using the Murray scale at day 3, 7, 14 and 28 after the administration of HCR040 | Day 28
  Murray scale from 0 to 4 where lower scores represent improvement
Vasopressor-free days 28 days after the administration of HCR040 | Day 28
ICU-free days 28 days after the administration of HCR040 | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Fermin Labayen Beraza, MD, Principal Investigator — Hospital de Cruces
Locations (2):
- Spain (2):
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Fundación Jiménez Díaz, Madrid